CLINICAL TRIAL: NCT00871559
Title: A Phase 1, Multiple-Dose Study of the Safety and Tolerability of Single Agent REGN421 Administered Every 2 or 3 Weeks in Patients With Advanced Solid Malignancies
Brief Title: A Multiple-Ascending-Dose Study of the Safety and Tolerability of REGN421(SAR153192) in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R421-ST-0804
Record Dates: First submitted 2009-03-25; First posted 2009-03-30 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Advanced Solid Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Q2W (Experimental): REGN421 (SAR153192) taken once every two weeks (Q2W)
  Interventions: Drug: REGN421(SAR153192)

INTERVENTIONS:
Drug: REGN421(SAR153192)

SUMMARY:
The purpose of this study is to assess the safety and tolerability of REGN421 (SAR153192) in patients with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older
2. Histologically diagnosis of advanced solid malignancy, with no standard therapeutic options of proven benefit.
3. Patients with measurable or non-measurable disease
4. At least 6 weeks must have elapsed since the last dose of bevacizumab (AvastinTM)
5. At least 4 weeks must have elapsed since the last major surgery
6. For women of childbearing potential, a negative urine pregnancy test at the screening visit
7. Willingness to use adequate contraception during the full course of the study. Systemic hormonal contraceptive agents are excluded
8. Willing, committed, and able to return for ALL clinic visits and complete all study-related procedures.
9. Able to read, understand and willing to sign the informed consent form

Exclusion Criteria:

1. Medical history of myocardial infarction or cardiomyopathy
2. Unstable angina
3. NYHA class II - IV congestive heart failure
4. Patients under treatment with more than 2 antihypertensive medications
5. History of bleeding peptic ulcer disease, erosive gastritis, intestinal perforation, or clinically significant GI hemorrhage within 6 months of study drug administration
6. Diabetic retinopathy
7. Patients requiring anticoagulation
8. Hypersensitivity to doxycycline or related compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 18 months

SECONDARY OUTCOMES:
Preliminary evidence of antitumor activity | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (8):
- United States (8):
  - Aurora, Colorado
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - New York, New York
  - Columbus, Ohio
  - Oklahoma City, Oklahoma